CLINICAL TRIAL: NCT05119569
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy of Fenebrutinib in Relapsing Multiple Sclerosis
Brief Title: A Study to Investigate the Efficacy of Fenebrutinib in Relapsing Multiple Sclerosis (RMS)
Acronym: FENopta
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN43271; 2021-003772-14 (EudraCT Number); 2022-502619-13-00 (EU CTIS Number)
Record Dates: First submitted 2021-10-29; First posted 2021-11-15 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — fenebrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor will also be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fenebrutinib (Experimental): Participants will receive oral fenebrutinib.
  Interventions: Drug: Fenebrutinib
- Placebo (Placebo Comparator): Participants will receive oral placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenebrutinib — Fenebrutinib will be administered orally.
  Arms: Fenebrutinib
Drug: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
This is a study evaluating the effect of fenebrutinib on brain magnetic resonance imaging (MRI) in participants with RMS. The safety and pharmacokinetics of fenebrutinib will also be evaluated. Participants will be randomized to receive either fenebrutinib or placebo. This study consists of two parts: Double-blind treatment (DBT) phase and an optional Open-label extension (OLE) phase.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RMS in accordance with the revised 2017 McDonald Criteria.
* Expanded Disability Status Scale (EDSS) score of 0 - 5.5 at screening.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating sperm.

Exclusion Criteria:

* Disease duration of > 10 years from the onset of symptoms and an EDSS score at screening < 2.0.
* Female participants who are pregnant or breastfeeding, or intending to become pregnant.
* Male participants who intend to father a child during the study.
* A diagnosis of Primary Progressive Multiple Sclerosis (PPMS) or non-active Secondary Progressive Multiple Sclerosis (SPMS).
* Any known or suspected active infection at screening, including but not limited to a positive screening tests for Hepatitis B and C, an active or latent or inadequately treated infection with tuberculosis (TB), a confirmed or suspected progressive multifocal leukoencephalopathy (PML).
* History of cancer including hematologic malignancy and solid tumors within 10 years of screening.
* Presence of other neurological disorders that could interfere with the diagnosis of MS or with the assessments of safety or efficacy during the study.
* Clinically significant cardiovascular, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic or gastrointestinal disease.
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
* History of alcohol or other drug abuse within 12 months prior to screening.
* History of or currently active primary or secondary (non-drug-related) immunodeficiency, including known history of HIV infection.
* Inability to complete an MRI scan.
* Adrenocorticotropic hormone or systemic corticosteroid therapy within 4 weeks prior to screening.
* Receipt of a live-attenuated vaccine within 6 weeks prior to randomization.
* Any previous treatment with immunomodulatory or immunosuppressive medication without an appropriate washout period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2026-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (2):
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Cleveland Clinic Lou Ruvo, Las Vegas, Nevada
- University Clinical Centre of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Croatia (4):
  - Clinical Hospital Center Rijeka - PPDS, Rijeka
  - General Hospital Varazdin, Varaždin
  - Klinicki bolnicki centar Zagreb, Zagreb
  - Poliklinika Solmed, Zagreb
- Czechia (4):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Vseobecna Fakultni Nemocnice V Praze - CRC - PPDS, Prague
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Clinical Hospital Centre Zemun, Zemun
- Univerzitna nemocnica Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Bar-Or A, Dufek M, Budincevic H, Drulovic J, Habek M, Hua LH, Weber MS, Thomas P, Napieralski J, Mitzner MC, Ratchford JN, Clayton D, Harp CT, Kuruvilla D, Qi Q, Chen YF, Xu Y, Goodyear A, Oh J; FENopta Study Group. Safety and efficacy of fenebrutinib in relapsing multiple sclerosis (FENopta): a multicentre, double-blind, randomised, placebo-controlled, phase 2 trial and open-label extension study. Lancet Neurol. 2025 Aug;24(8):656-666. doi: 10.1016/S1474-4422(25)00174-7. PMID 40683275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across 18 sites in 6 countries (Bosnia and Herzegovina, Croatia, Czech Republic, Serbia, Slovakia, and the United States). This study is still ongoing.
Pre-assignment Details: This study consists of two parts: Double-blind treatment (DBT) phase and an optional Open-label extension (OLE) phase. A total of 129 participants were screened, of which 109 were randomized into the fenebrutinib arm and placebo arm in a 2:1 ratio.
Groups:
- DBT Phase: Fenebrutinib: Participants received fenebrutinib, 200 milligrams (mg), orally, twice daily (BID) for 12 weeks during the DBT phase.
- DBT Phase: Placebo: Participants received fenebrutinib matching placebo, orally, BID for 12 weeks during the DBT phase.
- OLE Phase: Fenebrutinib From Fenebrutinib: Participants who received fenebrutinib in the DBT phase were given an option to receive fenebrutinib, 200 mg, orally, BID up to a maximum of 192 weeks in the OLE phase.
- OLE Phase: Fenebrutinib From Placebo: Participants who received fenebrutinib matching placebo in the DBT phase were given an option receive fenebrutinib, 200 mg, orally, BID up to a maximum of 192 weeks in the OLE phase.
Period: Double Blind Treatment Phase
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo | OLE Phase: Fenebrutinib From Fenebrutinib | OLE Phase: Fenebrutinib From Placebo
Started | 73 | 36 | 0 | 0
Completed | 65 | 34 | 0 | 0
Not Completed | 8 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0 | 0
Period: Open Label Extension Phase
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo | OLE Phase: Fenebrutinib From Fenebrutinib | OLE Phase: Fenebrutinib From Placebo
Started | 0 (Participants who completed the DBT Period were given the option to enroll in the OLE Period to receive fenebrutinib.) | 0 (Participants who completed the DBT Period were given the option to enroll in the OLE Period to receive fenebrutinib.) | 65 (65 participants who completed the DBT Period enrolled into the OLE Period.) | 34 (34 participants who completed the DBT Period enrolled into the OLE Period.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 65 | 34
Not completed — Ongoing in the study | 0 | 0 | 65 | 34

BASELINE CHARACTERISTICS:
Population: All Randomized Participants set included all randomized participants grouped by treatment as assigned by randomization.
Groups:
- DBT Phase: Fenebrutinib: Participants received fenebrutinib, 200 mg, orally, BID for 12 weeks during the DBT phase.
- Total: Total of all reporting groups
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo | Total
Number analyzed (Participants) | 73 | 36 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (8.5) | 39.8 (7.7) | 39.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 26 | 78
  Male | 21 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 72 | 36 | 108
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 73 | 36 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: DBT Phase: New Gadolinium (Gd) - Enhancing T1 Lesion Rate Observed on Magnetic Resonance Imaging (MRI) Scans of the Brain Over 12 Weeks
Description: Radiologic evaluation for Gd enhancing T1 lesion rate was performed using a standardized MRI protocol at screening, and at Weeks 4, 8, and 12. All MRI scans were read by a centralized reading center for efficacy endpoints. The total number of new Gd-enhancing T1 lesions were calculated as the sum of the individual number of new lesions observed at Weeks 4, 8 and 12. The lesion rate (new lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different number of scans.
Time Frame: MRI scans performed at Weeks 4, 8 and 12
Population: All Randomized Participants set included all randomized participants grouped by treatment as assigned by randomization. Overall number analyzed is the number of participants with evaluable post-baseline MRI scans.
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 70 | 36
adjusted number of new lesions per scan | 0.077 [0.043 to 0.135] | 0.245 [0.144 to 0.418]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.0022, Negative Binomial Regression Model; Rate Ratio = 0.313, 95% CI 2-sided [0.149 to 0.658]

2. Secondary Outcome: DBT Phase: New or Enlarging T2 - Weighted Lesion Rate Observed on MRI Scans of the Brain Over 12 Weeks
Description: Radiologic evaluation for new or enlarging T2 - weighted lesion rate was performed using a standardized MRI protocol at screening, and at Weeks 4, 8, and 12. All MRI scans were read by a centralized reading center for efficacy endpoints. Total number of new or enlarging T2-weighted lesions were calculated as the sum of the individual number of new or enlarging lesions at Weeks 4, 8, and 12. The lesion rate (new/enlarging lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different numbers of scans.
Time Frame: MRI scans performed at Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 70 | 36
adjusted number of new lesions per scan | 0.168 [0.102 to 0.277] | 0.634 [0.375 to 1.071]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.0004, Negative Binomial Regression Model; Rate Ratio = 0.265, 95% CI 2-sided [0.128 to 0.550]

3. Secondary Outcome: DBT Phase: Proportion of Participants Free From Any New Gd - Enhancing T1 Lesions and New or Enlarging T2 - Weighted Lesions Observed on MRI Scans of the Brain Over 12 Weeks
Description: Radiologic evaluation for new Gd - enhancing T1 lesion and new or enlarging T2 - weighted lesions were performed using a standardized MRI protocol at screening, and at Weeks 4, 8, and 12. All MRI scans were read by a centralized reading center for efficacy endpoints. The total number of new Gd-enhancing T1 lesions and new or enlarging T2 - weighted lesions were calculated as the sum of the individual number of lesions observed at Weeks 4, 8 and 12. Analysis was performed using a logistic regression model performed on the status of both new T1 Gd+ lesion and new or enlarging T2-weighted lesions post-baseline (present or not) adjusted for the stratification factor(s) presence or absence of T1 Gd+ lesions on the screening MRI.
Time Frame: MRI scans performed at Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 70 | 36
proportion of participants | 72.9 | 50.0
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.0117, Logistic Regression Model; Odds Ratio (OR) = 4.005, 95% CI 2-sided [1.317 to 13.078]

4. Secondary Outcome: DBT Phase: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity, is a congenital anomaly or birth defect.
Time Frame: Up to Week 12
Population: Safety population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 73 | 36
Participants
  AEs | 28 | 12
  SAEs | 0 | 0

5. Secondary Outcome: OLE Phase: Number of Participants With AEs and SAEs
Description: as for outcome 4
Time Frame: OLE Baseline (DBT Week 12) up to Week 192
Reporting Status: Not Posted, anticipated posting 2027-12

6. Secondary Outcome: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS=assessment tool used to assess lifetime suicidality of a participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, & attempts with actual/potential lethality. Categories have binary responses (yes/no) & include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher= suicidal ideation or behavior.
Time Frame: Up to Week 192
Reporting Status: Not Posted, anticipated posting 2027-12

7. Secondary Outcome: Plasma Concentrations of Fenebrutinib at Specified Timepoints
Time Frame: Up to Week 192
Reporting Status: Not Posted, anticipated posting 2027-12

8. Other Pre Specified Outcome: DBT Phase: New Gd - Enhancing T1 Lesion Rate Observed on MRI Scans of the Brain at Week 4
Description: Radiologic evaluation for Gd enhancing T1 lesion rate was performed using a standardized MRI protocol at screening, and at Week 4. All MRI scans were read by a centralized reading center for efficacy endpoints. The lesion rate (new lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different number of scans.
Time Frame: MRI scan performed at Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 70 | 36
adjusted number of new lesions per scan | 0.210 [0.115 to 0.382] | 0.269 [0.128 to 0.565]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.5889, Negative Binomial Regression Model; Rate Ratio = 0.780, 95% CI 2-sided [0.316 to 1.922]

9. Other Pre Specified Outcome: DBT Phase: New Gd - Enhancing T1 Lesion Rate Observed on MRI Scans of the Brain at Week 8
Description: Radiologic evaluation for Gd enhancing T1 lesion rate was performed using a standardized MRI protocol at screening, and at Week 8. All MRI scans were read by a centralized reading center for efficacy endpoints. The lesion rate (new lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different number of scans.
Time Frame: MRI scan performed at Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 67 | 34
adjusted number of new lesions per scan | 0.025 [0.006 to 0.101] | 0.325 [0.150 to 0.702]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.0011, Negative Binomial Regression Model; Rate Ratio = 0.076, 95% CI 2-sided [0.016 to 0.355]

10. Other Pre Specified Outcome: DBT Phase: New Gd - Enhancing T1 Lesion Rate Observed on MRI Scans of the Brain at Week 12
Description: Radiologic evaluation for Gd enhancing T1 lesion rate was performed using a standardized MRI protocol at screening, and at Week 12. All MRI scans were read by a centralized reading center for efficacy endpoints. The lesion rate (new lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different number of scans.
Time Frame: MRI scan performed at Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 63 | 33
adjusted number of new lesions per scan | 0.007 [0.001 to 0.052] | 0.066 [0.013 to 0.324]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.0038, Negative Binomial Regression Model; Rate Ratio = 0.104, 95% CI 2-sided [0.022 to 0.481]

11. Other Pre Specified Outcome: DBT Phase: New or Enlarging T2 - Weighted Lesion Rate Observed on MRI Scans of the Brain at Week 4
Description: Radiologic evaluation for new or enlarging T2 - weighted lesion rate was performed using a standardized MRI protocol at screening, and at Week 4. All MRI scans were read by a centralized reading center for efficacy endpoints. The lesion rate (new/enlarging lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different number of scans.
Time Frame: MRI scan performed at Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 70 | 36
adjusted number of new lesions per scan | 0.456 [0.274 to 0.757] | 0.891 [0.490 to 1.620]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.0958, Negative Binomial Regression Model; Rate Ratio = 0.512, 95% CI 2-sided [0.233 to 1.126]

12. Other Pre Specified Outcome: DBT Phase: New or Enlarging T2 - Weighted Lesion Rate Observed on MRI Scans of the Brain at Week 8
Description: Radiologic evaluation for new or enlarging T2 - weighted lesion rate was performed using a standardized MRI protocol at screening, and at Week 8. All MRI scans were read by a centralized reading center for efficacy endpoints. The lesion rate (new/enlarging lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different number of scans.
Time Frame: MRI scan performed at Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 67 | 34
adjusted number of new lesions per scan | 0.058 [0.023 to 0.144] | 0.549 [0.314 to 0.958]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p < 0.0001, Negative Binomial Regression Model; Rate Ratio = 0.105, 95% CI 2-sided [0.039 to 0.283]

13. Other Pre Specified Outcome: DBT Phase: New or Enlarging T2 - Weighted Lesion Rate Observed on MRI Scans of the Brain at Week 12
Description: Radiologic evaluation for new or enlarging T2 - weighted lesion rate was performed using a standardized MRI protocol at screening, and at Week 12. All MRI scans were read by a centralized reading center for efficacy endpoints. The lesion rate (new/enlarging lesions per scan) was estimated from a negative binomial regression model for the total number of events and was adjusted for the covariate 'presence or absence of T1 Gd+ lesions on the screening MRI'. Log-transformed number of scans were included in the negative binomial model as an "offset" variable to account for different number of scans.
Time Frame: MRI scan performed at Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted number of new lesions per scan
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
Number analyzed (Participants) | 63 | 33
adjusted number of new lesions per scan | 0.015 [0.003 to 0.068] | 0.282 [0.135 to 0.586]
Statistical Analysis 1: Comparison: DBT Phase: Fenebrutinib vs DBT Phase: Placebo; Test type: Superiority; p = 0.0001, Negative Binomial Regression Model; Rate Ratio = 0.053, 95% CI 2-sided [0.012 to 0.233]

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: Safety population included all participants who received any study drug. Data collected up to the primary completion date is reported here. Adverse events section will be updated one year after the study completion date.
Arm/Group | DBT Phase: Fenebrutinib | DBT Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/36
Other Adverse Events (participants affected / at risk) | 8/73 | 4/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBT Phase: Fenebrutinib (N=73) | DBT Phase: Placebo (N=36)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Hepatic enzyme abnormal (Investigations) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT05119569/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT05119569/SAP_001.pdf